CLINICAL TRIAL: NCT04587193
Title: Safety and Efficacy of State-of-the-Art Exoskeleton Technology to Improve Mobility in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented the study from being able to be completed
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20020066
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: Gait; Balance; Freezing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PD participants (Experimental): Subjects will participate in a total of 10 walking sessions, twice per week for 5 weeks, while wearing a robotic-assist gait training device. There will also be 3 additional visits for assessments at: baseline (up to 1 prior to treatment), post (1 week after last treatment), and final (4-6 weeks after last treatment).
  Interventions: Device: Robotic-assist gait training device

INTERVENTIONS:
Device: Robotic-assist gait training device — PD participants will walk while wearing a robotic-assist gait training device

SUMMARY:
The purpose of this study is to test the safety and efficacy of using of a portable exoskeleton for walking training in persons with Parkinson's disease that have gait mobility problems and/or postural instability.

DETAILED DESCRIPTION:
This is a feasibility study to examine a novel application of state-of-the-art robotic-assist gait training to improve mobility in people with Parkinson's disease (PD). The study will investigate the utility of the Keeogo® exoskeleton (a robotic-assist gait training device) for people with PD. The Keeogo® offers advantages of being lightweight and portable (for eventual home use) and is relatively quick to attach and remove. The aims here are to establish the safety of the Keeogo® for gait training in persons with PD and to preliminarily assess the potential efficacy of the Keeogo® for better balance control, gait mobility and fall reduction in persons with PD.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's Participant

1. age 21 years or older,
2. PD confirmed by a movement disorder specialist using UK Brain Bank Criteria,
3. H&Y stage II, III, IV, or V.

Caregiver participant

1. Caregiver of PD participant and is willing to complete questionnaire
2. moderate to severe cognitive impairment / dementia (Montreal Cognitive Assessment < 17/30) except in cases where the clinician and the participants Legally Authorized Representative both determine the participant can safely complete the study

Exclusion Criteria:

Parkinson's Participant

1. neurological, musculoskeletal, or other disorders unrelated to PD contributing to impairment of gait, stance, balance or coordination,
2. history of implantable cardiac device or ablative surgery,
3. moderate to severe cognitive impairment / dementia (Montreal Cognitive Assessment < 17/30),
4. uncontrolled orthostatic hypotension,
5. feeding tube or associated port placement (PEG/J-PEG),
6. body height less than 5'1" or greater than 6'3" and
7. body weight greater than 250 pounds.

Caregiver participant

1) Unwilling to complete questionnaire

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Baron, MD, Principal Investigator — Virginia Commonwealth University Health System; Robert Hand, PT, DPT, Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregiver Participants: Caregivers of persons enrolled in study (optional)
Period: Overall Study
Arm/Group | PD Participants | Caregiver Participants
Started | 6 | 2
Completed | 0 | 0
Not Completed | 6 | 2
Not completed — Screen failure after consent | 3 | 0
Not completed — Device broke during study | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Caregiver Participants: Participant's caregivers QOL will be assessed using the Parkinson's Disease Carer Questionnaire (PD-Carer), a 29 item measure of health related quality of life for use with carers of people with Parkinson's disease. Each item is scored from 0 to 4. Total scores are then added. Total scores range from 0 (no problem at all) to 116 (worst level of problem).
- Total: Total of all reporting groups
Arm/Group | PD Participants | Caregiver Participants | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Portable Exoskeleton
Description: Number of "prevented" or "near falls" requiring physical assistance by the investigative training team experienced by the participant during throughout the training.
Time Frame: At the end of treatment (5 weeks)
Measure: Number; unit: Number of prevented/near falls
Arm/Group | PD Participants
Number analyzed (Participants) | 3
Number of prevented/near falls | 0

2. Secondary Outcome: Change in Walking Capacity
Description: Walking capacity will be assessed using the 6-Minute Walking Test (6MWT) that assesses distance (in feet) walked to determine aerobic capacity and endurance. Participants will be asked to walk as far as possible in 6 minutes and the total distance will be recorded. The change in walking capacity from baseline to the week 5 treatment.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: Total distance (feet)
Arm/Group | PD Participants
Number analyzed (Participants) | 3
Total distance (feet)
  Baseline | 226 [181 to 262]
  After 4 treatments | 182 [125 to 239]

3. Secondary Outcome: Change in Freezing of Gait (FOG)
Description: FOG will be assessed using the 6MWT. FOG will be assess using 2 gait related questions on the Unified Parkinson's Disease Rating Scale (UPDRS). Scores are summed and range from 0 (normal) to 4 (very poor).
Time Frame: 6 weeks
Population: Only 1 participant performed study activities that collected this outcome measure.
Measure: Number; unit: Change in score
Arm/Group | PD Participants
Number analyzed (Participants) | 1
Change in score
  Baseline | 2
  1 wk post treatment | 4

4. Secondary Outcome: Change in Balance
Description: The Berg Balance Scale (BBS) assesses balance via asking the participant to perform 14 functional activities. Each functional activity is rated on a 5 point scale from 0 (unable) to 4 (able safety or with minimal aid). The score on each functional activity is then added to get an overall score from 0 to 56. Scores range from 0 to 56 with higher scores indicating better balance.
Time Frame: 6 weeks
Population: Only 1 participant performed study activities that collected this outcome measure.
Measure: Number; unit: score on scale
Arm/Group | PD Participants
Number analyzed (Participants) | 1
score on scale
  Baseline | 47
  1 wk post treatment | 52

5. Secondary Outcome: Change in Motor Symptoms
Description: The Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part IIIMDS-UPDRS, part III will be used to assess motor symptoms and fluctuations of Parkinson Disease (PD). This outcome measure will be used to report a change in PD motor symptoms from baseline. Scores range from 0 (best score) to 56 (worst score) with higher scores indicating more symptoms.
Time Frame: 6 weeks
Population: Only 1 participant performed study activities that collected this outcome measure.
Measure: Number; unit: Change in score
Arm/Group | PD Participants
Number analyzed (Participants) | 1
Change in score
  Baseline | 55
  1 wk post treatment | 45

6. Secondary Outcome: Change in Quality of Life (QOL)
Description: Parkinson's Disease Questionnaire (PDQ39) is a 39 item self-report questionnaire assessing how often patients experience difficulties across the 8 quality of life dimensions of functioning and well-being. Items are scored from 0 (never) to 4 (always). All items are then added to get a total score. Total scores can range from 0 to 156. The lower the total score, the better quality of life.
Time Frame: 6 weeks
Population: Only 1 participant performed study activities that collected this outcome measure.
Measure: Number; unit: Change in score
Arm/Group | PD Participants
Number analyzed (Participants) | 1
Change in score
  Baseline | 53
  1 wk post treatment | 34

7. Secondary Outcome: Change in Caregiver QOL
Description: Participant's caregivers QOL will be assessed using the Parkinson's Disease Carer Questionnaire (PD-Carer), a 29 item measure of health related quality of life for use with carers of people with Parkinson's disease. Each item is scored from 0 to 4. Total scores are then added. Total scores range from 0 (no problem at all) to 116 (worst level of problem).
Time Frame: 6 weeks
Population: Only 1 participant performed study activities that collected this outcome measure.
Measure: Number; unit: Change in score
Groups:
- Caregiver Participants: Subjects will be asked to complete the Parkinson's Disease Carer Questionnaire 3 times; once at the PD patient's screening visit, once at the PD patient's post-treatment visit and lastly are the PD patient's durability visit.
Arm/Group | Caregiver Participants
Number analyzed (Participants) | 1
Change in score
  Prescreen visit | 18
  Post-treatment visit | 22

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | PD Participants | Caregiver Participants
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD Participants (N=3) | Caregiver Participants (N=1)
Fatigue (General disorders) | 1 | NA
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04587193/Prot_002.pdf